CLINICAL TRIAL: NCT04718103
Title: A 52-week, Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-centre Study of the Efficacy and Safety of GSK3511294 Adjunctive Therapy in Adult and Adolescent Participants With Severe Uncontrolled Asthma With an Eosinophilic Phenotype
Brief Title: A Study of GSK3511294 (Depemokimab) in Participants With Severe Asthma With an Eosinophilic Phenotype
Acronym: SWIFT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213744
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: Asthma; Eosinophilic phenotype; Exacerbations; GSK3511294 (Depemokimab); Placebo
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to receive either GSK3511294 (Depemokimab) or placebo as an adjunct therapy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK3511294 (Experimental): Participants received a 100 milligram (mg) dose of GSK3511294 subcutaneous (SC) injection once every 26 weeks (week 0 and week 26). Participants were to be maintained on their existing baseline maintenance asthma standard of care (SOC) treatment throughout the study.
  Interventions: Biological: GSK3511294
- Placebo (Placebo Comparator): Participants received placebo SC injection once every 26 weeks (week 0 and week 26). Participants were to be maintained on their existing baseline maintenance asthma SOC treatment throughout the study.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK3511294 — GSK3511294 was administered using a pre-filled syringe.
  Other Names: Depemokimab
  Arms: GSK3511294
Biological: Placebo — Placebo was administered as normal saline using a pre-filled syringe.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of GSK3511294 (Depemokimab) as an adjunctive therapy in participants with severe uncontrolled asthma with an eosinophilic phenotype.

ELIGIBILITY:
Key inclusion criteria for study:

* Adults and adolescents greater than or equal to (>=)12 years of age, at the time of signing the informed consent/assent.
* Participants must have a documented physician diagnosis of asthma for >=2 years that meets the National Heart, Lung, and Blood Institute guidelines (NHLBI) or Global Initiative for Asthma (GINA) guidelines and

  1. Eosinophilic phenotype: participants who have, or with high likelihood of having, asthma with an eosinophilic phenotype as per randomization criteria, and
  2. Exacerbation history: participants who have previously confirmed history of >=2 exacerbations requiring treatment with systemic corticosteroid (CS) (Intramuscular [IM], Intravenous [IV], or oral), in the 12 months prior to Visit 1, despite the use of medium to high-dose ICS. For participants receiving maintenance CS, the CS treatment for the exacerbations must have been a two-fold dose increase or greater.
* Persistent airflow obstruction as indicated by (i) For participants >=18 years of age at Visit 1, a pre-bronchodilator FEV1 less than (<)80 percent (%) predicted National Health and Nutrition Examination Survey (NHANES III) recorded at Visit 1.

(ii) For participants 12-17 years of age at Visit 1: A pre-bronchodilator FEV1 <90% predicted (NHANES III) recorded at Visit 1 or FEV1: Forced Vital Capacity (FVC) ratio <0.8 recorded at Visit 1.

* A well-documented requirement for regular treatment with medium to high dose ICS (in the 12 months prior to Visit 1 with or without maintenance OCS). The maintenance ICS dose must be >=440 micrograms fluticasone propionate (FP) hydrofluoroalkane product (HFA) daily, or clinically comparable (GINA, 2020). Participants who are treated with medium dose ICS will also need to be treated with LABA to qualify for inclusion.
* Current treatment with at least one additional controller medication, besides ICS, for at least 3 months (for example [e.g.], LABA, LAMA, leukotriene receptor antagonist [LTRA], or theophylline).

Key inclusion criteria for randomization:

* An elevated peripheral blood eosinophil count of >=300 cells per microliter demonstrated in the past 12 months prior to Visit 1 that is related to asthma or an elevated peripheral blood eosinophil count of >=150 cells per microliter at Screening Visit 1 that is related to asthma.
* Evidence of airway reversibility or responsiveness as documented by either:

  (i) Airway reversibility (FEV1>=12% and 200 milliliter [mL]) demonstrated at Visit 1 or Visit 2 using the Maximum Post Bronchodilator Procedure or (ii) Airway reversibility (FEV1>=12% and 200 mL) documented in the 24 months prior to Visit 2 (randomization visit) or (iii) Airway hyper-responsiveness (methacholine: Provocative concentration causing a 20% fall in FEV1 [PC20] of <8 milligrams per milliliter (mg/mL), histamine: Provocative dose that decreases FEV1 by 20% [PD20] of <7.8 micromoles, mannitol: decrease in FEV1 as per the labelled product instructions) documented in the 24 months prior to Visit 2 (randomization visit).

Key exclusion criteria for study:

* Presence of a known pre-existing, clinically important lung condition other than asthma. This includes (but is not limited to) current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* Participants with other conditions that could lead to elevated eosinophils such as hyper-eosinophilic syndromes including (but not limited to) Eosinophilic Granulomatosis with Polyangiitis (EGPA, formerly known as Churg-Strauss Syndrome) or Eosinophilic Esophagitis.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to screening (Participants that had localized carcinoma of the skin which was resected for cure will not be excluded).
* Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* Participants who have known, pre-existing, clinically significant cardiac, endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, hematological or any other system abnormalities that are uncontrolled with standard treatment.
* Participants with current diagnosis of vasculitis. Participants with high clinical suspicion of vasculitis at screening will be evaluated and current vasculitis must be excluded prior to enrolment.
* Participants who have received mepolizumab (Nucala), reslizumab (Cinqair/Cinqaero), or benralizumab (Fasenra) within 12 months prior to Visit 1 or who have a previous documented failure with Anti-Interleukin-5/Anti-Interleukin-5 receptor (anti-IL-5/5R) therapy.
* Participants who have received omalizumab (Xolair) or dupilumab (Dupixent) within 130 days prior to Visit 1.
* Participants who have received any monoclonal antibody (mAb) within 5 half-lives of Visit 1.
* Previously participated in any study with mepolizumab, reslizumab, or benralizumab and received study intervention (including placebo) within 12 months prior to Visit 1.
* Corrected QT interval using Fridericia's formula (QTcF) >=450 milliseconds (msec) or QTcF >=480 msec for participants with Bundle Branch Block at screening Visit 1.
* Current smokers or former smokers with a smoking history of >=10 pack years (number of pack years = [number of cigarettes per day/ 20] multiplied by number of years smoked). A former smoker is defined as a participant who quit smoking at least 6 months prior to Visit 1.
* Participants with allergy/intolerance to the excipients of GSK3511294 or any mAb or biologic.

Key exclusion criteria for randomization:

* QTcF >= 450 msec or QTcF >=480 msec for participants with Bundle Branch Block, at randomization Visit 2 are excluded. Participants are excluded if an abnormal Electrocardiogram (ECG) finding from the 12-lead ECG conducted at Screening Visit 1 is considered to be clinically significant and would impact the participant's participation during the study, based on the evaluation of the Investigator.
* Participants with a clinically significant asthma exacerbation in the 7 days prior to randomization should have their randomization visit delayed until the investigator considers the participant's asthma to be stable.
* Any changes in the dose or regimen of Baseline ICS and/or additional controller medication (except for treatment of an exacerbation) during the run-in period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (108):
- United States (37):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Lancaster, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Lafayette, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Northfield, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Edmond, Oklahoma
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, DuBois, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Allen, Texas
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (2):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, South Brisbane, Queensland
- Canada (5):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Kamloops, British Columbia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Windsor
- Czechia (3):
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Teplice
- France (6):
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
- Hungary (3):
  - GSK Investigational Site, GOdOll?
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Szigetvár
- Italy (10):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Foggia
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Monserrato CA
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pietra Ligure SV
  - GSK Investigational Site, Rozzano MI
  - GSK Investigational Site, Salerno
  - GSK Investigational Site, Siena
  - GSK Investigational Site, Tradate VA
- Japan (17):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Poland (6):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Strzelce Opolskie
  - GSK Investigational Site, Wroclaw
- Spain (14):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, La Laguna Santa Cruz
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Linkou - Taoyuan Hsien
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Jackson DJ, Wechsler ME, Jackson DJ, Bernstein D, Korn S, Pfeffer PE, Chen R, Saito J, de Luiz Martinez G, Dymek L, Jacques L, Bird N, Schalkwijk S, Smith D, Howarth P, Pavord ID; SWIFT-1 and SWIFT-2 Investigators; SWIFT-1 Investigators; SWIFT-2 Investigators. Twice-Yearly Depemokimab in Severe Asthma with an Eosinophilic Phenotype. N Engl J Med. 2024 Dec 19;391(24):2337-2349. doi: 10.1056/NEJMoa2406673. Epub 2024 Sep 9. PMID 39248309
- [Derived] Jackson DJ, Bourdin A, Blackorby A, Leslie A, Vichiendilokkul A, Howarth P, Karkoszka N, Fujieda S, Cornet M. Safety and Tolerability of Twice-Yearly Depemokimab in Patients with Asthma and Chronic Rhinosinusitis with Nasal Polyps: Pooled Results from SWIFT-1/-2 and ANCHOR-1/-2. Adv Ther. 2025 Dec 29. doi: 10.1007/s12325-025-03457-4. Online ahead of print. PMID 41461999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 397 participants were randomized to the study. Of which 380 participants were included in Full analysis set (FAS) population. FAS included all randomized participants who received at least 1 dose of study intervention excluding 12 participants from 2 sites with Good Clinical Practice (GCP) violation. Five (5) participants were randomized in error and did not receive any study drug.
Pre-assignment Details: A total of 397 were randomized in the study.
Period: Overall Study
Arm/Group | GSK3511294 | Placebo
Started (Randomized) | 263 | 134
Full Analysis Population | 252 | 128
Completed | 233 | 117
Not Completed | 30 | 17
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 4 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Randomized, not treated | 4 | 1
Not completed — GCP violations | 7 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set population included all randomized participants who received at least one dose of study intervention excluding participants from 2 sites with GCP violation. Participants were analyzed according to the intervention they were allocated at randomization.
Groups:
- GSK3511294: Participants received a 100 mg dose of GSK3511294 SC injection once every 26 weeks (week 0 and week 26). Participants were to be maintained on their existing baseline maintenance asthma SOC treatment throughout the study.
- Total: Total of all reporting groups
Arm/Group | GSK3511294 | Placebo | Total
Number analyzed (Participants) | 252 | 128 | 380
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 53.6 (16.00) | 51.2 (16.58) | 52.8 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 81 | 241
  Male | 92 | 47 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into 'Others' category to minimize the possibility of re-identification of participants.
  Participants
    Asian | 52 | 23 | 75
    White | 181 | 91 | 272
    Others | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Clinically Significant Exacerbations up to 52 Weeks
Description: Clinically significant exacerbations recorded were defined as worsening of asthma requiring the use of systemic corticosteroids (CS) [such as intramuscular (IM), intravenous (IV) or oral] and/or hospitalization and/or Emergency Department (ED) visit. For all participants, IV or oral steroids (e.g., prednisone) for at least 3 days or a single IM corticosteroid dose is required. For participants on maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days is required. Exacerbations recorded in the electronic case report form (eCRF) were considered as verified clinically significant exacerbations and included in the primary analysis. Exacerbations separated by less than 7 days was treated as a continuation of the same exacerbation.
Time Frame: Up to Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbation per participant per year
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 252 | 128
Exacerbation per participant per year | 0.56 [0.44 to 0.70] | 1.08 [0.83 to 1.41]
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; To demonstrate the superiority of GSK3511294 100 mg SC + SoC following two doses (at Week 0 and at Week 26) compared with placebo + SoC, assessed by the annualized rate of clinically significant exacerbations measured over the study intervention period of 52 weeks; Test type: Superiority — Analysis performed using a generalized linear model assuming a negative binomial distribution and covariates of treatment group, baseline ICS dose (medium or high), exacerbation history (2, 3, 4+), geographical region and baseline pre-bronchodilator percent predicted Forced Expiratory Volume in one second (FEV1) and offset of log (total time in the study in years); p < 0.001, Negative Binomial Distribution; Rate Ratio = 0.52, 95% CI 2-sided [0.36 to 0.73]

2. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: The SGRQ is a 50-item patient-reported outcome tool used to measure Quality of Life in participants with airway obstruction diseases. The questions are designed to be self-completed by the participant. The total score was calculated by the symptom score, activity and impact score; and summarizing the impact of the disease on overall health status on 0-100 rating scale. Scores are expressed as a percentage of overall impairment where 100 representing worst possible health status and 0 indicating best possible health status. Higher scores indicating greater impairment of quality of life. Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline (Day 1) and Week 52
Population: The FAS included all randomized participants who received at least 1 dose of study intervention excluding participants from 2 sites with GCP violation. Participants were analyzed according to the intervention they were allocated at randomization. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 246 | 124
Scores on a scale | -14.80 (1.041) | -12.49 (1.455)
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; To demonstrate the superiority of GSK3511294 100 mg SC + SoC following two doses (at Week 0 and at Week 26) compared with placebo + SoC, assessed by SGRQ Total Score measured over the study intervention period of 52 weeks; Test type: Superiority; p = 0.200, Mixed Models Repeated Measures (MMRM); Least-square (LS) means = -2.31, 95% CI 2-sided [-5.84 to 1.23]

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score at Week 52
Description: The ACQ-5 is a five-item questionnaire developed as a measure of participants asthma symptom control. The questions are designed to be self-completed by the participant. The 5 questions enquired to recall how their asthma had been during the previous week and to respond about the frequency and/or severity of symptoms (nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheezing). The overall ACQ-5 response option is the mean score of all 5 questions representing 0 with no impairment/limitation and 6 as total impairment/ limitation. Higher scores indicated more limitations and lower score with better asthma control. Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 246 | 124
Scores on a scale | -0.81 (0.065) | -0.70 (0.091)
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; Analysis performed using a repeated measures model with covariates of treatment group, baseline ICS dose (medium or high), exacerbation history (2, 3, 4+), geographical region, baseline ACQ-5 score, baseline pre-bronchodilator percent predicted FEV1, visit, visit by baseline ACQ-5 score and visit by treatment group; Test type: Superiority; p = 0.333, Mixed Models Repeated Measures (MMRM); Difference in Least-Square Mean = -0.11, 95% CI 2-sided [-0.33 to 0.11]

4. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in One Second (FEV1) At Week 52
Description: Forced Expiratory Volume in One Second (FEV1) is defined as the volume of air that can be forced out in one second after taking a deep breath by a person and will be measured by spirometry testing. Change from Baseline in clinic pre-bronchodilator FEV1 was determined. Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 239 | 119
Liters (L) | 0.240 (0.0286) | 0.184 (0.0407)
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; Analysis performed using a repeated measures model with covariates of treatment group, baseline ICS dose (medium or high), exacerbation history (2, 3, 4+), geographical region, baseline pre-bronchodilator FEV1, visit, visit by baseline pre-bronchodilator FEV1 and visit by treatment group; Test type: Superiority; p = 0.267, Mixed Models Repeated Measures (MMRM); Difference in Least-Square Means = 0.056, 95% CI 2-sided [-0.043 to 0.154]

5. Secondary Outcome: Change From Baseline in Asthma Nighttime Symptom Diary (ANSD) Weekly Mean Score at Week 52
Description: The ANSD is a 6-item self-administered patient reported diary developed by Patient Related Outcomes (PRO) Consortium's Asthma Working Group to facilitate comprehensive and reliable assessment of asthma symptoms from a participant's perspective. Participants were required to rate the severity of symptoms in 3 core categories: breathing symptoms (wheezing, shortness of breath), chest symptoms (chest tightness, chest pain) and cough. The ANSD was to be completed before going to bed and refers to asthma symptoms during the day. Symptoms are rated at their worst using an 11-point numeric rating scale ranging from 0 (None) to 10 (As bad as you can imagine). Higher scores indicate more severe symptoms. Mean daily scores of ANSD was calculated by weekly intervals. The baseline values were defined as the average score from Day -7 to Day -1 inclusive (at least 4 days must be non-missing). Change from Baseline was defined as value at each time point minus Baseline value.
Time Frame: Baseline to Week 52
Population: All participants in the FAS population (excluding participants from 2 sites with GCP violation) for whom at least one ANSD questionnaire was administered. Participants were analyzed according to the intervention they were allocated at randomization. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 232 | 117
Scores on a scale | -1.18 (0.091) | -0.97 (0.127)
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; Analysis performed using a repeated measures model with covariates of treatment group, baseline ICS dose (medium or high), exacerbation history (2, 3, 4+), geographical region, baseline ANSD weekly mean score, baseline pre-bronchodilator percent predicted FEV1, visit, visit by baseline ANSD weekly mean score and visit by treatment group; Test type: Superiority; p = 0.173, Mixed Models Repeated Measures (MMRM); Difference in Least square means = -0.21, 95% CI 2-sided [-0.52 to 0.09]

6. Secondary Outcome: Change From Baseline in Asthma Daily Symptom Diary (ADSD) Weekly Mean Score at Week 52
Description: The ADSD is a 6-item self-administered patient reported diary developed by patient related outcomes (PRO) Consortium's Asthma Working Group to facilitate comprehensive and reliable assessment of asthma symptoms from a participant's perspective. Participants were required to rate the severity of symptoms in 3 core categories: breathing symptoms (wheezing, shortness of breath), chest symptoms (chest tightness, chest pain) and cough. The ADSD was to be completed upon waking and refers to asthma symptoms during the night-time. Symptoms are rated at their worst using an 11-point numeric rating scale ranging from 0 (None) to 10 (As bad as you can imagine). Higher scores indicate more severe symptoms. Mean daily scores of ADSD was calculated by weekly intervals. The baseline values were defined as the average score from Day -7 to Day -1 inclusive (at least 4 days must be non-missing). Change from Baseline was defined as value at each time point minus Baseline value.
Time Frame: Baseline to Week 52
Population: All participants in the FAS population (excluding participants from 2 sites with GCP violation) for whom at least one ADSD questionnaire was administered. Participants were analyzed according to the intervention they were allocated at randomization. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 249 | 126
Scores on a scale | -1.13 (0.080) | -0.93 (0.112)
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; Analysis performed using a repeated measures model with covariates of treatment group, baseline ICS dose (medium or high), exacerbation history (2, 3, 4+), geographical region, baseline ADSD weekly mean score, baseline pre-bronchodilator percent predicted FEV1, visit, visit by baseline ADSD weekly mean score and visit by treatment group; Test type: Superiority; p = 0.138, Mixed Models Repeated Measures (MMRM); Difference in Least square means = -0.21, 95% CI 2-sided [-0.48 to 0.07]

7. Secondary Outcome: Annualized Rate of Exacerbations Requiring Hospitalization and/or Emergency Department (ED) Visit up to 52 Weeks
Description: Annualized Rate of exacerbations of asthma were defined as worsening of asthma which required use of systemic corticosteroids (CSs) and/or hospitalization and/or Emergency Department (ED) visit. For all participants, IV or oral steroids (e.g., prednisone) for at least 3 days or a single IM CS dose is required. For participants on maintenance systemic CSs, at least double the existing maintenance dose for at least 3 days is required. Exacerbations separated by less than 7 days will be treated as a continuation of the same exacerbation. Exacerbations Requiring Hospitalization and/or ED Visit are reported here.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbation per participant per year
Arm/Group | GSK3511294 | Placebo
Number analyzed (Participants) | 252 | 128
Exacerbation per participant per year | 0.05 [0.02 to 0.09] | 0.11 [0.05 to 0.22]
Statistical Analysis 1: Comparison: GSK3511294 vs Placebo; Test type: Superiority — Analysis performed using a generalized linear model assuming a negative binomial distribution and covariates of treatment group, baseline ICS dose (medium or high), exacerbation history (2, 3, 4+), geographical region and baseline pre-bronchodilator percent predicted FEV1; p = 0.087, Negative binomial distribution; Rate Ratio = 0.42, 95% CI 2-sided [0.16 to 1.13]

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected from the start of the study intervention (Day 1) till follow up week 56.
Description: All-cause mortality, SAEs and Non-SAEs were reported for the Safety Population which included all randomized participants who received at least 1 dose of study treatment excluding participants from 2 site with GCP violation. AEs were reported treatment-wise. One participant was randomized to receive GSK3511294 but received one dose of placebo in error and did not receive the second planned dose. This participant was included in the actual treatment group (placebo) for the safety population.
Arm/Group | GSK3511294 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/129
Serious Adverse Events (participants affected / at risk) | 19/251 | 13/129
Other Adverse Events (participants affected / at risk) | 138/251 | 80/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3511294 (N=251) | Placebo (N=129)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase abnormal (Investigations) | 1 (1) | 0 (0)
Blood bilirubin abnormal (Investigations) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 6 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3511294 (N=251) | Placebo (N=129)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 12 (12) | 10 (11)
COVID-19 (Infections and infestations) | 36 (38) | 19 (20)
Influenza (Infections and infestations) | 5 (5) | 9 (9)
Lower respiratory tract infection (Infections and infestations) | 4 (5) | 5 (8)
Nasopharyngitis (Infections and infestations) | 33 (45) | 27 (44)
Pharyngitis (Infections and infestations) | 10 (10) | 1 (1)
Respiratory tract infection (Infections and infestations) | 5 (7) | 4 (4)
Rhinitis (Infections and infestations) | 7 (7) | 5 (6)
Sinusitis (Infections and infestations) | 11 (11) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 21 (29) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (8) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (7)
Dizziness (Nervous system disorders) | 8 (10) | 1 (1)
Headache (Nervous system disorders) | 20 (30) | 10 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 3 (3)
Hypertension (Vascular disorders) | 6 (7) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT04718103/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04718103/SAP_001.pdf